CLINICAL TRIAL: NCT00147420
Title: RCT of Zhi Byed 11 (ZB11) Versus Misoprostol in Tibet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); University of Utah (Other); Health Bureau Tibet Autonomous Region (Unknown); University of California, San Francisco (Other); One Heart Project (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GN 10
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Hemorrhage
Keywords: Tibet; Third Stage Labor; Post Partum Hemorrhage; Misoprostol; Zhi Byed 11; Global Network
MeSH Terms: conditions — Hemorrhage; Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Zhi Byed 11

SUMMARY:
Previous research has confirmed that hemorrhage is among the most commonly encountered pregnancy complications in the Tibet Autonomous Region (TAR). This trial will test the effectiveness of a traditional Tibetan drug (Zhi Byed 11) vs. misoprostol to prevent postpartum hemorrhage (PPH) among women delivering vaginally in three hospitals in Lhasa, TAR.

DETAILED DESCRIPTION:
Post-partum hemorrhage (PPH) is one of the main direct causes of maternal mortality, particularly in rural areas with low access to skilled providers, blood banks, and surgical facilities. In addition to the mortality, PPH also accounts for a great number of morbidities, including anemia, renal and pulmonary problems, fatigue, and decreased resistance to infection, all major health problems affecting women in the TAR. Clinical research is rare in the Tibetan Autonomous Region (TAR) of the People's Republic of China. This trial will estimate the effect of prophylactic oral ZB 11 administered at the beginning of the second stage of labor versus prophylactic oral misoprostol, administered in the third stage of labor, in reducing the incidence of postpartum hemorrhage (defined as a measured blood loss of > 500 cc).

An observational postpartum blood measurement study was conducted. This included data collection on deliveries in three TAR hospital in Lhasa, piloting of consent forms and data collection instruments, and training in the use of a plastic drape for the measurement of postpartum blood loss.

This randomized, double masked trial will test the hypothesis that misoprostol is more effective than ZB11 in reducing the frequency of postpartum hemorrhage (defined as either a measured blood loss of > 500cc or administration of open label uterotonics within the one hour observation period after delivery).

An original sample of 848 women was increased and 967 consenting women were randomized (1:1) to a ZB11 or misoprostol arm. Since ZB 11 and misoprostol must be administered at different times, participants will receive either active ZB 11 or corresponding placebo at full dilation and active misoprostol or corresponding placebo immediately following the birth of the baby. The effectiveness of the study drug will be estimated by the postpartum blood loss that will be measured on all enrolled women with a blood collection drape.

ELIGIBILITY:
Inclusion and Exclusion Criteria

Adult, pregnant women who satisfy all the following criteria may be enrolled in the study. Pregnant women:

* who are delivering during the study period at one of the three hospitals
* who are 18 years of age or older at the time of delivery
* who are 28 weeks or more pregnant
* who are likely to have a normal vaginal delivery
* with singleton intrauterine pregnancy with vertex presentation either in early labor or in anticipation of induction of labor, and
* whose fetus is alive (has a heart rate >100bpm) at the time of screening
* who are able to give informed consent.

Any of the following criteria will exclude a woman from study participation:

* pre-term labor (<28 weeks)
* previous or planned cesarean delivery
* current multiple gestations
* active hemorrhaging
* severe anemia (Hgh <7)
* hypertension (persistent BP>140/90 or greater OR hypertension requiring treatment) [this criteria was omitted mid-study]
* maternal history of bleeding disorders
* known allergies to any medications (severe chronic allergic conditions)
* body temperature greater than 38ºC
* asthma (asthma requiring treatment)
* mental disability
* unable to focus on consent process due to imminent delivery

To be eligible for participation as a care provider, the participant must satisfy the following criteria:

* obstetrical care provider to pregnant woman in the study
* at least 18 years of age
* must be a physician or nurse midwife

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 848
Dates: Start 2005-09; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Postpartum hemorrhage
Maternal death

SECONDARY OUTCOMES:
Estimated average blood loss of women during birth

CONTACTS AND LOCATIONS:
Overall Officials: Michael Varner, MD, Principal Investigator — University of Utah
Locations (3):
- China (3):
  - Lhasa Maternal-Child Health (MCH) Hospital, Lhasa
  - Lhasa Municipal Hospital, Lhasa
  - The Mentzikhang Traditional Tibetan Medicine and Astrology Hospital, Lhasa

REFERENCES:
- See also: Global Network for Women and Children's Health Research — http://gn.rti.org
- See also: Research Triangle Institute International — http://www.rti.org